CLINICAL TRIAL: NCT07265830
Title: The Building Adaptive School-based Interventions for Caries Study (BASICS): A Phase III Sequential, Multiple-Assignment, Randomized Trial of Minimally Invasive Therapies to Reduce Treatment Nonresponse
Brief Title: Building Adaptive School-based Interventions for Caries
Acronym: BASICS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: i24-01908; R01MD019938 (NIH)
Record Dates: First submitted 2025-11-20; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries
Keywords: Dental caries; Adaptive interventions; Prevention; Child; Dynamic treatment regimes; SMART
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: BASICS is a phase-III Sequential, Multiple-Assignment, Randomized Trial (SMART)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Subgroup A, SDF only (Experimental): Single intervention: Silver diamine fluoride (SDF)
  Interventions: Device: Silver Diamine Fluoride (38%)
- Subgroup D, Sealant only (Active Comparator): Single intervention: Glass Ionomer Cement (GIC) Sealant
  Interventions: Device: Glass Ionomer Sealant
- Subgroup B, SDF + FV + Hygiene Intervention (Experimental): Nonresponse arm: SDF (First stage) + [SDF + Fluoride Varnish (FV) + Hygiene Intervention (Second Stage)]
  Interventions: Device: Silver Diamine Fluoride (38%); Device: Fluoride Varnishes; Behavioral: Hygiene Intervention
- Subgroup C, SDF + SMART + Sealant (Experimental): Nonresponse arm: SDF (First Stage) + [Silver Modified Atraumatic Restorative Treatment (SMART) + Sealant (Second Stage)]
  Interventions: Device: Silver Diamine Fluoride (38%); Device: Glass Ionomer Sealant
- Subgroup E, Sealant + SMART + FV + Hygiene Intervention (Experimental): Nonresponse arm: GIC Sealant (First Stage) + [ART + FV + Hygiene Intervention (Second Stage)]
  Interventions: Device: Glass Ionomer Sealant; Device: Fluoride Varnishes; Behavioral: Hygiene Intervention
- Subgroup F, Sealant + SMART (Experimental): Nonresponse arm: GIC Sealant (First Stage) + [SMART (Second Stage)]
  Interventions: Device: Silver Diamine Fluoride (38%); Device: Glass Ionomer Sealant

INTERVENTIONS:
Device: Silver Diamine Fluoride (38%) — Topically applied silver diamine fluoride 38% solution
  Arms: Subgroup A, SDF only; Subgroup B, SDF + FV + Hygiene Intervention; Subgroup C, SDF + SMART + Sealant; Subgroup F, Sealant + SMART
Device: Glass Ionomer Sealant — GIC Dental Sealants
  Arms: Subgroup C, SDF + SMART + Sealant; Subgroup D, Sealant only; Subgroup E, Sealant + SMART + FV + Hygiene Intervention; Subgroup F, Sealant + SMART
Device: Fluoride Varnishes — Topically applied fluoride varnish (FV)
  Arms: Subgroup B, SDF + FV + Hygiene Intervention; Subgroup E, Sealant + SMART + FV + Hygiene Intervention
Behavioral: Hygiene Intervention — Behavioral intervention to improve dental hygiene
  Arms: Subgroup B, SDF + FV + Hygiene Intervention; Subgroup E, Sealant + SMART + FV + Hygiene Intervention

SUMMARY:
Dental caries (tooth decay) is the world's most prevalent noncommunicable disease. Current preventive and therapeutic treatments are available that can be provided in a school-based health service environment. However, not all children respond to care, and school programs can result in under- or over-treatment, leaving children at high risk. The Building Adaptive School-based Interventions for Caries (BASICS) study will identify the optimal sequence and intensity of these treatments to minimize nonresponse, creating adaptive interventions tailored to specific needs in order to personalize school-based dental medicine.

DETAILED DESCRIPTION:
Dental caries is the world's most prevalent noncommunicable disease, with considerable health disparities found in low-income rural white children and low-income urban Hispanic/Latino and black children. To combat this silent epidemic, school-based caries prevention can increase access to critical dental care, reducing caries risk and mitigating its severe health and socioemotional consequences. However, despite the use of evidence-based interventions, approximately 30% of children participating in school-based caries prevention fail to respond to treatment ("nonresponse"), developing new caries and remaining at high risk for subsequent complications. Additionally, the sustainability of school-based prevention is jeopardized due to prohibitive costs, limitations of the professional workforce, and relying on treatments that are not optimized for individual patient needs. The Building Adaptive School-based Interventions for Caries (BASICS) study will develop and assess personalized, resource-efficient approaches to school caries prevention using adaptive interventions. Evaluated by embedding dynamic treatment regimes (DTR) within a Sequential, Multiple-Assignment, Randomized Trial (SMART) design, investigators will explore a number of hypotheses related to adaptive preventive interventions for caries. First, investigators will test the effects of adaptive interventions on reducing treatment nonresponse using generalized linear mixed models, followed by identifying the best dynamic treatment regime using augmented inverse probability weighted marginal structural models for causal effect estimation. Investigators will subsequently build an optimal adaptive intervention using Q-learning, tailoring treatments to individual patient attributes and responsiveness. Investigators will conclude with a microcosting analysis of the adaptive interventions, ultimately quantifying the intervention costs under different implementation scenarios and taking the first step towards understanding how much payers should reimburse for adaptive interventions. Successful completion of this project will produce resource-efficient adaptive prevention interventions (API) to reduce treatment nonresponse and improve oral health.

ELIGIBILITY:
Inclusion Criteria:

1. Be enrolled in participating schools
2. Be between the ages of 5 and 13 years
3. Provide parental/guardian informed consent
4. Child assent

Exclusion Criteria:

1. Ulcerative gingivitis or stomatitis
2. Known sensitivity to silver or other heavy-metal ions
3. More than six affected sites
4. Those who have had full mouth gingivectomies
5. Patients showing abnormal skin sensitization in daily circumstances
6. Those who have had pulp capping

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Dental Caries Incidence | Biannual assessment from enrollment to end of treatment (2.5 years)
  Number of teeth presenting with new caries
Caries Prevalence | Biannual assessment from enrollment to end of treatment (2.5 years)
  The prevalence of study participants with dental caries

CONTACTS AND LOCATIONS:
Overall Officials: Ryan R Ruff, PhD, MPH, Principal Investigator — New York University College of Dentistry/Epidemiology

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and de-identified patient data will be made available upon reasonable request and approval of a data use agreement.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting information will be available at the end of the trial for five years.
Access Criteria: Anyone with an approved data use agreement.

DOCUMENTS (2):
  • Study Protocol (2025-10-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT07265830/Prot_000.pdf
  • Informed Consent Form (2025-10-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT07265830/ICF_001.pdf